CLINICAL TRIAL: NCT00755300
Title: Total Knee Arthroplasty And Thromboembolism: A Comparison Between Two Surgical Techniques
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Amrik Singh, M.D., University of California Davis Department of Anesthesiology & Pain Medicine
Other Study IDs: 200614481
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Total Knee Replacement; Venous Thromboembolism
Keywords: Total knee replacement; esophageal echocardiography
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Standard Total Knee Replacement
  Interventions: Procedure: Measurement of total thrombolic load
- 2: Computer Guided Knee Replacement
  Interventions: Procedure: Measurement of total thrombolic load

INTERVENTIONS:
Procedure: Measurement of total thrombolic load — A video recording of the right atrium using TE echo will be used to quantitate the total thromboembolic load

SUMMARY:
In patients undergoing total knee arthroplasty, thromboembolism is a common occurrence, especially following tourniquet deflation. The resulting cardiopulmonary emboli can potentially lead to hypoxemia, hypotension, hemodynamic collapse and post operative cognitive dysfunction due to emboli. The standard surgical technique involves placing an intramedullary rod in the femur to determine the angle and degree of resection from the end of the femur. A new surgical technique utilizes computer navigation system to perform the desired cuts in the appropriate position. The investigators hypothesize that the avoidance of intramedullary instrumentation in computer assisted total knee replacement will result in fewer thromboembolic events compared with the standard technique using manual instrumentation in the femur. The present study will test this hypothesis by quantifying the extent of thromboembolism during both surgical techniques.

DETAILED DESCRIPTION:
Currently, Transesophageal Echocardiography (TEE) is routinely used intraoperatively to monitor patients undergoing total knee arthroplasty for thromboembolic events. Video recording (without any patient identifiers) of the TEE loops before and after tourniquet release, offline analysis to quantify the extent of thromboembolism and the two surgical techniques will be compared. Patients are assigned to a particular technique according to some non-rigid criteria. This study has no impact on their selection into one group or the other. Participation in this study does not influence the choice/selection. We will simply record and analyze the echo loops in twenty patients already assigned to each surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo Total Knee Arthroplasty at UC Davis Medical Center
* 18 years and above

Exclusion Criteria:

* Any contraindication to perform TEE

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Total venous embolic load | Acute, 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amrik Singh, M.D., Principal Investigator — Associate Professor, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States